CLINICAL TRIAL: NCT00630708
Title: Safety of Dual Blockage of Rennin-angiotensin System in Patients With Advanced Renal Insufficiency
Acronym: SDBRAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant differences observed between groups.
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nanfang200803
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Renal insufficiency; Benazepril; Losartan; combination treatment; Safety
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — benazepril; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Benazepril group
  Interventions: Drug: Benazepril
- 2 (Active Comparator): Losartan group
  Interventions: Drug: Losartan
- 3 (Active Comparator): Benazepril+Losartan group
  Interventions: Drug: Benazepril+Losartan

INTERVENTIONS:
Drug: Benazepril — 20 mg per day
  Other Names: Lotensin
  Arms: 1
Drug: Losartan — 100 mg per day
  Other Names: Cozaar
  Arms: 2
Drug: Benazepril+Losartan — combination treatment of 10 mg benazepril and 50 mg losartan per day
  Other Names: Lotensin+Cozaar
  Arms: 3

SUMMARY:
The primary aim of the present study is to assess the safety of combined treatment of benazepril (an ACE inhibitor) or losartan (an ARB) in non-diabetic patients with advanced renal insufficiency.

DETAILED DESCRIPTION:
Interruption of the renin-angiotensin systerm (RAS) with an angiotensin-converting enzyme (ACE) inhibitor or an angiotensin II receptor blocker (ARB) slows the progression of chronic renal insufficiency in the presence or absence of diabetes. Even for advanced chronic renal insufficiency (stage 4 CKD), ACE inhibitors and ARBs can still provide renoprotection. Some clinical studies showed that dual RAS blockage seemed to enhance the antiproteinuric effect compared with single-agent ACE inhibitor or ARB and then improve renal survival. However, in the only one randomized controlled trial investigating the renoprotection of combined ACE inhibitor and ARB for mild or moderate chronic renal insufficiency (the mean creatinine value is 2.9mg/dl), the incidence of hyperkalemia was increased in combination therapy compared with monotherapy. Although increase of hyperkalemia was not statistical significant, it suggested that combination treatment of ACEI and ARB might increase the incidence of hyperkalemia in patients with advanced renal insufficiency. However, it is still undetermined whether combination treatment of ACE inhibitor and ARB is safe as an ACE inhibitor or ARB monotherapy in advanced non-diabetic chronic renal insufficiency (stage 4 CKD). The primary aim of the present study is to assess the safety of combined treatment of benazepril (an ACE inhibitor) or losartan (an ARB) in non-diabetic patients with advanced renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Serum creatinine concentration of 3.0 to 5.0 mg per deciliter (265 to 442 µmol/L)
2. Creatinine clearance of 15 to 30 ml per minute per 1.73m2, with variations of less than 30 percent in the three months before screening evaluation
3. non-diabetic renal disease
4. Persistent heavier proteinuria (defined by urinary protein excretion of more than 0.3g per day for three or more months without evidence of urinary tract infection or overt heart failure [a New York Heart Association class of Ⅲ or Ⅳ])
5. had not received ACE inhibitors or ARBs for at least two weeks before screening

Exclusion Criteria:

1. No history of allergic reaction to drugs, especially ACE inhibitors and/or ARBs
2. Hyper-or hypokalemia (serum potassium concentration 5.6 mmol per liter or more，or 3.5 mmol per liter or less)
3. Malignant hypertension (blood pressure >180/120 mm Hg) or blood pressure <110mm Hg without antihypertensive treatment
4. Treatment with drugs affecting serum potassium such as diuretic, β2 receptor blocker et al.
5. Treatment with corticosteroids, non-steroidal anti-inflammatory drugs, or immunosuppressive drugs, especially ciclosporin A
6. Myocardial infarction or cerebrovascular accident in the year preceding the trial
7. Nephrotic syndrome (albuminaemia less than 25 g/L)
8. Renovascular disease or connective-tissue disease
9. Obstructive uropathy
10. Immediate need for dialysis
11. Pregnancy or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2008-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with increase in serum potassium ≥6.0 mmol/L. | Every 4 weeks

SECONDARY OUTCOMES:
The proportion of patients with serum creatinine increase >30% | Every 4 weeks
The proportion of patients with drug-related cough | Every 4 weeks
The proportion of patients with hopotension (systolic blood pressure <110 mmHg despite withdrawal of all additional antihypertensive medication) | Every 4 weeks
The proportion of patients with non-fatal cardiovascular events | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fan Fan Hou, M.D.,Ph.D., Principal Investigator — Renal Division, Nanfang Hospital,Southern Medical University
Locations (1):
- Renal Division, Nanfang Hospital,Southern Medical University, Guangzhou, Guangdong, China